CLINICAL TRIAL: NCT03495908
Title: Efficacy and Safety Comparison Between U-100 Regular Human Insulin and Rapid Acting Insulin When Delivered by VGo Wearable Insulin Delivery in Type 2 Diabetes
Brief Title: Regular Insulin vs Rapid Insulin Delivered by V-Go
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Coast Institute for Research (Network)
Collaborators: Valeritas, Inc. (Industry); Dallas Diabetes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGo Switch
Record Dates: First submitted 2018-03-17; First posted 2018-04-12 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus
Keywords: VGo; Insulin; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VGo with Regular Human Insulin (Experimental): U-100 short-acting insulin, Regular, human insulin rDNA origin, including Humulin® R, Novolin® R, and ReliOn (Novolin R) delivered by V-Go
  Interventions: Device: VGo
- VGo with Rapid Acting Insulin (Active Comparator): U-100 fast-acting insulin including Humalog® (insulin lispro, rDNA origin) or NovoLog® (insulin aspart, rDNA origin), which have both been tested by Valeritas, Inc. and found to be safe for use in the V-Go or Apidra® (insulin glulisine, rDNA origin) delivered by V-Go
  Interventions: Device: VGo

INTERVENTIONS:
Device: VGo — Eligible subjects will be randomized to either stay on RAI delivered by V-Go or randomized to switch to U-100 RHI delivered by V-Go.

SUMMARY:
The purpose of the study is to collect data about how well U-100 Regular Human Insulin can be used in the V-Go Insulin Delivery Device compared to U-100 Rapid Acting Insulin in the V-Go Insulin Delivery Device. The data collected will be used to see how much subjects' blood sugar levels change over time after they switch from using U-100 Rapid Acting Insulin to U-100 Regular Human Insulin within their V-Go Insulin Delivery Device.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years at time of study enrollment
2. Diagnosed with T2D for at least 6 months prior to screening
3. Screening visit A1C ≥ 7.0% and ≤ 12.5%
4. Prescribed a stable (less than 20% change in the past 30 days) of rapid acting U-100 insulin delivered via V-Go insulin delivery device
5. Ability to read and understand English
6. Willing to complete all study related activities
7. Willing and able to understand and sign a written ICF indicating that they agree to participate and have been informed of all pertinent aspects of the study
8. Must be willing to take and record 7 glucose measurements per time period (pre-morning meal (fasting), pre-midday meal, pre-evening meal, and 2-hours after the start of the morning, midday, and evening meals, and at bedtime) three times throughout the study (prior to Visit 2, 3, and 4).
9. Completed a 7-point glucose profile prior to Visit 2
10. Able (by insurance or financial means) to cover the initial investment and ongoing cost of the V-Go insulin delivery device, insulin (current rapid acting insulin or potential new regular human insulin), personal glucometer and supplies for the length of the study.

Exclusion Criteria:

1. Subject with confirmed Type 1 diabetes
2. More than 1 episode of severe hypoglycemia (defined as requiring third party assistance) within 3 months of study entry
3. History of hypoglycemia unawareness
4. Require supplemental insulin in addition to V-Go therapy
5. Woman of child-bearing potential who has a positive pregnancy test at screening or plans to become pregnant during the course of the study. Women of childbearing potential are defined as any female who has experienced menarche and who it NOT permanently sterile of postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without and alternative medical cause.
6. Woman who are lactating.
7. Use of any oral, injectable, or IV steroids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study
8. A recipient of a solid organ transplant
9. Current use of U-100 RHI in V-Go within 90 days of screening
10. Current use of U-500 RHI in V-Go within 90 days of screening
11. Currently on dialysis
12. Medical or other problems which in the opinion of the investigator will render study participation unsafe.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Macon, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mora PF, Sutton DR, Gore A, Baliga B, Goldfaden RF, Nikkel C, Sink Ii J, Adams-Huet B. Efficacy, safety and cost-effectiveness comparison between U-100 human regular insulin and rapid acting insulin when delivered by V-Go wearable insulin delivery device in type 2 diabetes. BMJ Open Diabetes Res Care. 2020 Nov;8(2):e001832. doi: 10.1136/bmjdrc-2020-001832. PMID 33214190

RESULTS

PARTICIPANT FLOW:
Groups:
- VGo With Regular Human Insulin: Switch to U-100 Regular Human Insulin (RHI) delivered by the V-Go insulin delivery device.
- VGo With Rapid Acting Insulin: Continue on U-100 Rapid Acting Insulin (RAI) delivered by the V-Go insulin delivery device.
Period: Overall Study
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Started | 69 | 67
Completed | 59 | 54
Not Completed | 10 | 13
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Physician Decision | 5 | 4
Not completed — No documented reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin | Total
Number analyzed (Participants) | 69 | 67 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 42 | 83
  >=65 years | 28 | 25 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.9) | 60.2 (11.6) | 61.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 43 | 82
  Male | 30 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 67 | 65 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 30 | 50
  White | 47 | 35 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 69 | 67 | 136
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of Hemoglobin A1c] | 8.5 (1.4) | 8.5 (1.5) | 8.5 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Change In HbA1c Between Groups After 12 Weeks of Treatment. Non-inferiority Hypothesis.
Description: Per protocol population for assessment of non-inferiority of RHI. Week 12 change from baseline in HbA1c comparison of RHI versus RAI estimated treatment difference.
Time Frame: Baseline and Week 12
Population: Per protocol
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 59 | 54
percent | -0.5966 [-0.9041 to -0.2892] | -0.3759 [-0.6973 to -0.05455]
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; RHI - RAI estimated treatment difference (ETD) in HbA1c. Per-protocol analysis is the pre-specified primary outcome; Test type: Non-Inferiority — Non-inferiority margin is 0.4% HbA1c; p = 0.007, Mixed Models Analysis — Non-inferiority p-value based on the 0.4% non-inferiority margin; Mean Difference (Net) = -0.2207, 95% CI 2-sided [-0.6654 to 0.2241] — RHI - RAI estimated treatment difference. Upper confidence interval 0.22 is less than the 0.4% non-inferiority margin

2. Secondary Outcome: Evaluate the Prevalence of Hypoglycemic Events Between Groups Based on 7- Point Glucose Profiles.
Description: Number of participants reporting 7-Point Hypoglycemia based on 7-point glucose profiles. Intent-to-treat (ITT) Population N=136
Time Frame: Baseline and Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 69 | 67
Participants
  Pre-randomization | 9 | 8
  Post-randomization | 11 | 12
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; Post-randomization prevalence of hypoglycemia based on 7-point glucose profiles; Test type: Superiority — Comparison of Post-randomization prevalence of hypoglycemia based on 7-point glucose profiles; p = .82, Fisher Exact

3. Secondary Outcome: Evaluate the Incidence of Hypoglycemic Events Between Groups Based on 7- Point Glucose Profiles.
Description: Level 1 (≤70 mg/dL or (<3.9 mmol/L)) and level 2 hypoglycemia (<54 mg/dL (<3.0 mmol/L)) events are analyzed. No level 3 events were reported for either group.
Time Frame: Baseline and Week 12
Population: Intent-to-treat safety population, n=136
Measure: Number; unit: Events per person weeks
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 69 | 67
Events per person weeks
  Pre-randomization | 0.069 | 0.065
  Post-randomization | 0.016 | 0.017
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; Level 1 (≤70 mg/dL or (<3.9 mmol/L)) and level 2 hypoglycemia (<54 mg/dL (<3.0 mmol/L)) events are analyzed. No level 3 events were reported for either group; Test type: Superiority — Analysis of the 7-point profiles within the ITT population (n=136); p = 0.861, Regression, Poisson — Results are from a Poisson regression model with repeated measures; generalized estimating equations (GEE) approach; Poisson regression model with repeated measures; generalized estimating equations (GEE) approach; Risk Ratio (RR) = 0.925, 95% CI 2-sided [0.386 to 2.217] — The incidence rate ratio quantitates the risk of hypoglycemia in the RHI group (RR numerator) compared with the RAI group (RR numerator). Results from Poisson regression model with repeated measures; generalized estimating equations (GEE) approach

4. Secondary Outcome: Evaluate the Change in Total Daily Doses (Units/kg) of Insulin Between Groups After 12 Weeks of Treatment.
Description: Between group differences in Insulin TDD U/day. Intent-to-treat Population, n=136
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: units/kg
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 69 | 67
units/kg
  Baseline TDD U/kg | 0.65 [0.61 to 0.69] | 0.65 [0.61 to 0.69]
  End of study TDD U/kg | 0.66 [0.62 to 0.70] | 0.67 [0.61 to 0.71]
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; RHI versus RAI for Insulin Intent-to-treat Population N=136 Mixed Model Estimates for Insulin TDD U/kg I; Test type: Superiority; p = 0.415, Mixed Models Analysis; Mean Difference (Net) = -0.01073, 95% CI 2-sided [-0.03674 to 0.01528] — Between Group Comparison (RHI-RAI) Estimated Treatment Difference (ETD) mixed effects model analysis

5. Secondary Outcome: Evaluate the Change in Total Daily Doses (TDD), Units/Day of Insulin Between Groups After 12 Weeks of Treatment.
Description: RHI versus RAI, comparing the change in total daily dose (TDD), units/day of insulin between groups. Intent-to-treat Population N=136
Time Frame: Baseline and Week 12
Population: Intent-to-treat Population N=136
Measure: Least Squares Mean (95% Confidence Interval); unit: units/day
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 69 | 67
units/day
  Baseline Insulin TDD, U/day | 61.13 [57.66 to 64.60] | 60.90 [57.37 to 64.42]
  End of Study Insulin TDD, U/day | 61.90 [58.38 to 65.41] | 62.74 [59.15 to 66.32]
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; Test type: Superiority; p = 0.320, Mixed Models Analysis; Mean Difference (Net) = -1.0776, 95% CI 2-sided [-3.2139 to 1.0587] — Between Group Comparison (RHI-RAI) Estimated Treatment Difference (ETD) mixed effects model analysis

6. Secondary Outcome: Evaluate the Difference in Direct Pharmacy Insulin Costs to Insurance Payor Using Wholesale Acquisition Costs Between Groups.
Description: Cost Analysis for direct diabetes-related pharmacy insulin costs. All insulin costs are normalized to 30-days and based on the prescribed TDD at V2 (Baseline) and at study end (EOS) and multiplying the insulin dose in units by the average unit cost of the prescribed insulin
Time Frame: Baseline and Week 12
Population: Per-protocol population, n=113
Measure: Mean (Standard Deviation); unit: US dollar
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 59 | 54
US dollar
  Baseline Insulin Cost, $ | 515.68 (123.01) | 518.31 (124.23)
  End of Study Insulin Cost, $ | 265.19 (61.39) | 533.66 (118.51)
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -265.85, 95% CI 2-sided [-288.60 to -243.11] — Estimated Treatment Difference (RHI-RAI) from repeated measures mixed model least squares estimates

7. Secondary Outcome: Evaluate the Change In HbA1c Between Groups After 12 Weeks of Treatment. Intent-to-treat Population Secondary Outcome, Non-inferiority Hypothesis.
Description: Intent-to-treat population secondary outcome for assessment of non-inferiority of RHI. Week 12 change from baseline in HbA1c comparison of RHI versus RAI estimated treatment difference.
Time Frame: Baseline and Week 12
Population: Intent-to-treat secondary outcome of HbA1c response for assessment of non-inferiority of RHI compared to RAI
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of Hemoglobin A1c
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
Number analyzed (Participants) | 69 | 67
percentage of Hemoglobin A1c | -0.5484 [-0.8618 to -0.2349] | -0.4167 [-0.7425 to -0.09088]
Statistical Analysis 1: Comparison: VGo With Regular Human Insulin vs VGo With Rapid Acting Insulin; Intent-to-treat secondary outcome of HbA1c response for assessment of non-inferiority of RHI compared to RAI; Test type: Non-Inferiority — Change in A1C Non-inferiority Margin is 0.4%; p = 0.02, Mixed Models Analysis — p-value for non-inferiority; Mean Difference (Net) = -0.1317, 95% CI 2-sided [-0.5838 to 0.3205] — Between Group Difference (RHI-RAI) mixed effects repeated measures model analysis.Upper confidence interval 0.32 is less than the 0.4% non-inferiority margin

8. Other Pre Specified Outcome: Evaluate the Change in Glucose Patterns Between Groups Based on 7-point Glucose Profiles.
Description: Evaluate the change between baseline and week 12 in glucose patterns between groups based on 7-point glucose profiles.
Time Frame: Baseline and Week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks. From randomization to end of study.
Arm/Group | VGo With Regular Human Insulin | VGo With Rapid Acting Insulin
All-Cause Mortality (participants affected / at risk) | 1/69 | 0/67
Serious Adverse Events (participants affected / at risk) | 5/69 | 3/67
Other Adverse Events (participants affected / at risk) | 1/69 | 2/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VGo With Regular Human Insulin (N=69) | VGo With Rapid Acting Insulin (N=67)
Heart Attack (Cardiac disorders) | 0 (0) | 1 (1)
Wound (Infections and infestations) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening of A-fib (Cardiac disorders) | 1 (1) | 0 (0)
Bilateral Papillary Carcinoma (Endocrine disorders) | 1 (1) | 0 (0)
Worsening of CHF (Cardiac disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VGo With Regular Human Insulin (N=69) | VGo With Rapid Acting Insulin (N=67)
Upset stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) — Possibly related
Skin irritation, welt (Product Issues) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03495908/Prot_SAP_000.pdf